CLINICAL TRIAL: NCT01842997
Title: A Stratified and Controlled Clinical Trial With Split-virion, Non-adjuvanted Influenza A/H1N1 Vaccines in Healthy Pregnant Women
Brief Title: Safety of H1N1 Influenza Vaccination in Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Principal Investigator, fubaoma, prof., Jiangsu Province Centers for Disease Control and Prevention
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSEPI-001
Record Dates: First submitted 2013-04-24; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Virus Diseases; Respiratory Tract Infections; Influenza; Orthomyxoviridae Infections
Keywords: Flu; non-adjuvanted H1N1 vaccine; Safety; pregnant women
MeSH Terms: conditions — Virus Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- split-virion, non-adjuvanted H1N1 vaccine of 15 μg (Experimental): split-virion, non-adjuvanted H1N1 vaccine of 15 μg made by Shanghai Institute of Biological Products lot number: 200909008
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg

INTERVENTIONS:
Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg — 122 participants (19 at 5-9 weeks pregnant,36 at 10-19 weeks pregnant,13 at 20-29 weeks pregnant,54 at more than 30 weeks pregnant) received split-virion, non-adjuvanted H1N1 vaccine of 15 μg.

SUMMARY:
Since October 2009, H1N1 influenza vaccine has developed and approved of immunization in population in China. However, there was little epidemiological evidence of safety when vaccinated in healthy pregnant women. The main objective of this study is to assess the safety of split-virion inactivated H1N1 vaccine without adjuvant when administered in healthy pregnant women. It is a stratified and controlled clinical trial in healthy pregnant women. And participants were included up to 226 healthy pregnant women aged 18 -35 years old who have no history of novel influenza H1N1 infection or novel influenza H1N1 vaccination. The pregnancy week ranged from 5 weeks to 32 weeks. Subjects were divided into 2 groups: vaccinated group（122） and unvaccinated group（104）. Subjects in the vaccinated group were administered one dose of 15μg H1N1 vaccine. Subjects in the unvaccinated group received no vaccine as controls. Safety will be measured by assessment of pregnancy outcomes. And observation time for pregnancy outcomes was lasting for 28 days postpartum since vaccinated; and protective effect was observed for six months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women
2. Be able to show legal identity card for the sake of recruitment
3. Be able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
3. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
4. Autoimmune disease or immunodeficiency
5. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
6. Diabetes mellitus (type I or II), with the exception of gestational diabetes
7. History of thyroidectomy or thyroid disease that required medication within the past 12 months
8. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
9. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
10. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
11. History of any blood products or seasonal influenza vaccine administration within 3 months before the dosing
12. Administration of any other investigational research agents within 30 days before the dosing
13. Administration of any live attenuated vaccine within 30 days before the dosing
14. Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
15. Axillary temperature > 37.0 centigrade at the time of dosing
16. Psychiatric condition that precludes compliance with the protocol
17. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse Pregnancy Outcomes | 0-28 days postpartum
  include the following indicators： incidence of spontaneous abortion, incidence of induced abortion，incidence of Preterm, incidence of post-term pregnancy, proportion of underweight-Babies

SECONDARY OUTCOMES:
incidence of influenza-like illness | 0-6months

CONTACTS AND LOCATIONS:
Overall Officials: Fubao Ma, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention
Locations (1):
- Xiangshui Center for Disease Control and Prevention, Xiangshui, Jiangsu, China

REFERENCES:
- [Derived] Ma F, Zhang L, Jiang R, Zhang J, Wang H, Gao X, Li X, Liu Y. Prospective cohort study of the safety of an influenza A(H1N1) vaccine in pregnant Chinese women. Clin Vaccine Immunol. 2014 Sep;21(9):1282-7. doi: 10.1128/CVI.00375-14. Epub 2014 Jul 2. PMID 24990911